CLINICAL TRIAL: NCT03621696
Title: Phase II Trial of Surgery Followed by Risk-Directed Post-Operative Adjuvant Therapy for HPV-Related Oropharynx Squamous Cell Carcinoma: "The Minimalist Trial (MINT)"
Brief Title: Surgery Followed by Risk-Directed Post-Operative Adjuvant Therapy for HPV-Related Oropharynx Squamous Cell Carcinoma: "The Minimalist Trial (MINT)"
Acronym: MINT
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 201808045
Record Dates: First submitted 2018-07-26; First posted 2018-08-08 (Actual); Results first posted 2022-03-11 (Actual); Last update posted 2025-08-17 (Actual); Status verified 2025-08

CONDITIONS: HPV Related Oropharyngeal Squamous Cell Carcinoma
MeSH Terms: interventions — Cisplatin; Radiotherapy, Intensity-Modulated; Surgical Procedures, Operative

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- Arm 1: POAmCRT (Experimental): * Patients with extracapsular extension (ECE) or positive margin but not clinical or pathologic T4 or clinical N3 disease
  * Standard of care surgery (surgical resection of the primary tumor via a transoral approach and surgical management of cervical lymph nodes
  * Treated with post-operative adjuvant modified chemoradiation therapy (POAmCRT) which is 42 Gy radiation therapy in 21 doses and 1 dose of cisplatin.
  * It is recommended that radiation therapy begin within 28-49 days (no later than 56 days) after surgical resection
  * Intensity modulated radiation therapy (IMRT) or intensity modulated proton therapy (IMPT) is to be used for this study
  Interventions: Drug: Cisplatin; Radiation: Intensity modulated radiation therapy; Radiation: Intensity modulated proton therapy; Procedure: Surgery; Other: FACT-H&N; Other: MD Anderson Dysphagia Inventory; Other: University of Michigan Xerostomia Index; Other: Scale of Subjective Total Taste Acuity; Other: Neck Dissection Impairment Index
- Arm 2: POAmRT (Experimental): * Patients with no extracapsular extension (ECE) and no positive margins and not clinical or pathologic T4 or clinical N3 disease
  * Standard of care surgery (surgical resection of the primary tumor via a transoral approach and surgical management of cervical lymph nodes
  * Treated with post-operative adjuvant modified radiation therapy (POAmRT) which is 42 Gy radiation therapy in 21 doses
  * It is recommended that radiation therapy begin within 28-49 days (no later than 56 days) after surgical resection
  * Intensity modulated radiation therapy (IMRT) or intensity modulated proton therapy (IMPT) is to be used for this study
  Interventions: Radiation: Intensity modulated radiation therapy; Radiation: Intensity modulated proton therapy; Procedure: Surgery; Other: FACT-H&N; Other: MD Anderson Dysphagia Inventory; Other: University of Michigan Xerostomia Index; Other: Scale of Subjective Total Taste Acuity; Other: Neck Dissection Impairment Index
- Arm 3: POACRT (Experimental): * Patients with clinical or pathologic T4 or clinical N3 disease
  * Standard of care surgery (surgical resection of the primary tumor via a transoral approach and surgical management of cervical lymph nodes
  * Treated with post-operative adjuvant chemoradiation therapy (POACRT) which is 60 Gy radiation therapy in 30 doses and 3 doses of cisplatin (if there is pathologic evidence of ECE or positive margins)
  * The first dose of cisplatin will given on one of the days during the initial 5 days of radiation therapy, the 2nd dose on the day of radiation dose 16, and the 3rd dose on the day of radiation dose 26.
  * It is recommended that radiation therapy begin within 28-49 days (no later than 56 days) after surgical resection
  * Intensity modulated radiation therapy (IMRT) or intensity modulated proton therapy (IMPT) is to be used for this study
  Interventions: Drug: Cisplatin; Radiation: Intensity modulated radiation therapy; Radiation: Intensity modulated proton therapy; Procedure: Surgery; Other: FACT-H&N; Other: MD Anderson Dysphagia Inventory; Other: University of Michigan Xerostomia Index; Other: Scale of Subjective Total Taste Acuity; Other: Neck Dissection Impairment Index

INTERVENTIONS:
Drug: Cisplatin — -100 mg/m^2 intravenous push bolus (IVPB)
  Other Names: Platinol®; Platinol-AQ®
  Arms: Arm 1: POAmCRT; Arm 3: POACRT
Radiation: Intensity modulated radiation therapy — -IMRT or IMPT can be used
  Other Names: IMRT
Radiation: Intensity modulated proton therapy — -IMRT or IMPT can be used
  Other Names: IMPT
Procedure: Surgery — -Standard of care
Other: FACT-H&N — -Baseline, interim assessment (14-42 days post-surgery), day 1 of radiation, day 21 of radiation, day 36 of radiation, 6 weeks after completion of adjuvant therapy, 4 months after the completion of adjuvant therapy, 6 months after the completion of adjuvant therapy, 12 months after the completion of adjuvant therapy, and 24 months after completion of adjuvant therapy
Other: MD Anderson Dysphagia Inventory — -Baseline, interim assessment (14-42 days post-surgery), day 1 of radiation, day 21 of radiation, day 36 of radiation, 6 weeks after completion of adjuvant therapy, 4 months after the completion of adjuvant therapy, 6 months after the completion of adjuvant therapy, 12 months after the completion of adjuvant therapy, and 24 months after completion of adjuvant therapy
Other: University of Michigan Xerostomia Index — -Baseline, interim assessment (14-42 days post-surgery), day 1 of radiation, day 21 of radiation, day 36 of radiation, 6 weeks after completion of adjuvant therapy, 4 months after the completion of adjuvant therapy, 6 months after the completion of adjuvant therapy, 12 months after the completion of adjuvant therapy, and 24 months after completion of adjuvant therapy
Other: Scale of Subjective Total Taste Acuity — -Baseline, interim assessment (14-42 days post-surgery), day 1 of radiation, day 21 of radiation, day 36 of radiation, 6 weeks after completion of adjuvant therapy, 4 months after the completion of adjuvant therapy, 6 months after the completion of adjuvant therapy, 12 months after the completion of adjuvant therapy, and 24 months after completion of adjuvant therapy
Other: Neck Dissection Impairment Index — -Baseline, interim assessment (14-42 days post-surgery), day 1 of radiation, day 21 of radiation, day 36 of radiation, 6 weeks after completion of adjuvant therapy, 4 months after the completion of adjuvant therapy, 6 months after the completion of adjuvant therapy, 12 months after the completion of adjuvant therapy, and 24 months after completion of adjuvant therapy

SUMMARY:
The overarching goal of the MINT trial is to reduce treatment-related toxicity while maintaining efficacy. Patients with HPV-related oropharyngeal squamous cell carcinoma (OPSCC) will undergo resection of the primary tumor site and involved/at risk regional neck nodes.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed HPV-related stages I-III OPSCC (8th edition of AJCC/UICC Staging Manual) or HPV-related neck node with unknown primary. HPV-related may be defined by p16 IHC stain and/or HPV-ISH or PCR using standard definitions of positive and negative test results.
* Primary tumor that will be resected via a transoral oral approach (conventional surgery, transoral laser microsurgery, transoral robotic surgery)
* Eastern Cooperative Oncology Group (ECOG) Performance Status (PS) 0-2.
* Normal organ and marrow function defined as:

  * Creatinine clearance > 50 cc/min.
  * ANC > 1,000/mcL.
  * Platelet count >100,000/mcL.
* At least 18 years of age.
* Women of childbearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control, abstinence) prior to study entry and for the duration of participation. Should a woman become pregnant or suspect she is pregnant while participating in this study, she must inform her treating physician immediately.
* Patient (or legally authorized representative) must be able to understand and willing to sign a written informed consent document.

Exclusion Criteria:

* Prior curative therapy for HNSCC.
* Patient must not have known distant metastatic disease at presentation.
* History of prior invasive malignancy diagnosed within 2 years prior to study enrollment; exceptions are malignancies with a low risk of metastasis or death (e.g., expected 5-year overall survival (OS) > 90%) that were treated with an expected curative outcome, such as squamous cell carcinoma of the skin, in-situ carcinoma of the cervix uteri, non-melanomatous skin cancer, carcinoma in situ of the breast, or incidental histological finding of prostate cancer (TNM stage of T1a or T1b).
* Receiving any other investigational agents.
* Uncontrolled serious inter-current illness or serious psychiatric illness/social situations that would limit compliance with study requirements.
* Pregnant and/or breastfeeding. A negative serum or urine pregnancy test is required at screening for all female patients of childbearing potential.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 63 (Actual)
Dates: Start 2018-10-23 (Actual); Primary Completion 2021-03-10 (Actual); Study Completion 2026-03-10 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Douglas Adkins, M.D., Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Alvin J. Siteman Cancer Center at Barnes-Jewish Hospital and Washington University School of Medicine — http://www.siteman.wustl.edu

RESULTS

PARTICIPANT FLOW:
Groups:
- Not Assigned to an Arm: -Patients were enrolled to the study but deemed ineligible to start treatment and were not enrolled to any arm.
Period: Overall Study
Arm/Group | Arm 1: POAmCRT | Arm 2: POAmRT | Arm 3: POACRT | Not Assigned to an Arm
Started | 21 | 31 | 6 | 5
Completed | 20 | 30 | 4 | 0
Not Completed | 1 | 1 | 2 | 5
Not completed — Not eligible | 0 | 0 | 0 | 5
Not completed — Withdrawal by Subject | 1 | 1 | 1 | 0
Not completed — Physician Decision | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm 1: POAmCRT | Arm 2: POAmRT | Arm 3: POACRT | Not Assigned to an Arm | Total
Number analyzed (Participants) | 21 | 31 | 6 | 5 | 63
Age, Continuous [Median (Full Range); unit: years] | 56 [37 to 72] | 58 [34 to 72] | 60 [51 to 63] | 57 [49 to 69] | 58 [34 to 72]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 4 | 0 | 0 | 5
  Male | 20 | 27 | 6 | 5 | 58
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 0 | 0 | 1
  Not Hispanic or Latino | 20 | 30 | 6 | 5 | 61
  Unknown or Not Reported | 0 | 1 | 0 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 2 | 0 | 1 | 0 | 3
  White | 19 | 31 | 5 | 5 | 60
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 21 | 31 | 6 | 5 | 63

OUTCOME MEASURES:

1. Primary Outcome: Mean Percent Weight Change
Description: * Weight in kilograms will be collected weekly during radiation
  * The percent weight loss from the baseline is calculated at any post-baseline
Time Frame: Starting at Day 1 and ending on the last day of radiation therapy (approximately 4 weeks)
Population: 1 participant not evaluable in Arm 2 and 2 participants not evaluable in Arm 3 as they didn't receive CRT.
Measure: Mean (95% Confidence Interval); unit: percent of change
Arm/Group | Arm 1: POAmCRT | Arm 2: POAmRT | Arm 3: POACRT
Number analyzed (Participants) | 20 | 30 | 4
percent of change | -4.89 [-6.24 to -3.54] | -3.18 [-4.19 to -2.17] | -10.11 [-15.79 to -4.43]

2. Secondary Outcome: Proportion of PEG Tube Placements in Each Arm
Description: -95% confidence intervals will be calculated assuming a binomial distribution
Time Frame: Through completion of follow-up (approximately 63 months)
Reporting Status: Not Posted

3. Secondary Outcome: Change in Serum Creatinine
Time Frame: Baseline to 6 weeks after POAmCRT (approximately 90 days)
Population: 1 participant not evaluable in Arm 2 and 2 participants not evaluable in Arm 3 as they didn't receive CRT.
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Arm 1: POAmCRT | Arm 2: POAmRT | Arm 3: POACRT
Number analyzed (Participants) | 21 | 30 | 4
mg/dL | 0.03 (0.09) | 0.08 (0.22) | -0.19 (0.19)

4. Secondary Outcome: Percentage of Participants Taking Narcotics
Description: -95% confidence intervals will be calculated assuming a binomial distribution
Time Frame: 6 weeks after POAmCRT (approximately 90 days)
Population: 1 participant not evaluable in Arm 2 and 2 participants not evaluable in Arm 3 as they didn't receive CRT.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Arm 1: POAmCRT | Arm 2: POAmRT | Arm 3: POACRT
Number analyzed (Participants) | 20 | 30 | 4
percentage of participants | 40 [16.5 to 63.5] | 20 [4.8 to 35.2] | 75 [54.6 to 100]

5. Secondary Outcome: Disease Recurrence Rate
Time Frame: 24 months post-treatment (approximately 27 months)
Measure: Count of Participants; unit: Participants
Arm/Group | Arm 1: POAmCRT | Arm 2: POAmRT | Arm 3: POACRT
Number analyzed (Participants) | 20 | 30 | 4
Participants | 2 | 1 | 3

6. Secondary Outcome: Progression-free Survival (PFS)
Time Frame: Through completion of follow-up (approximately 63 months)
Reporting Status: Not Posted

7. Secondary Outcome: Overall Survival (OS)
Time Frame: Through completion of follow-up (approximately 63 months)
Reporting Status: Not Posted

8. Other Pre Specified Outcome: Comparison of Quality of Life as Measured by the Neck Dissection Impairment Index
Description: -10-item self-administered questionnaire, which was designed to assess "quality of life related to shoulder dysfunction" after neck dissection. A 5-point response option (1 to 5) is provided for each item, with 1 being the most disability and 5 the least disability. The responses for all 10 items are added together to produce a raw score, which is then transformed to a score of 100 maximum. Higher scores represent less disability.
  --Captured at baseline, interim assessment (14-42 days post-surgery), Day 1 of radiation, Day 21 after start of radiation, Day 36 after start of radiation, and 6 weeks/4 months/6 months/12 months after completion of adjuvant therapy
Time Frame: From baseline through one year after completion of treatment (approximately 15 months)
Reporting Status: Not Posted

9. Other Pre Specified Outcome: Comparison of Quality of Life as Measured by the Scale of Subjective Total Taste Acuity
Description: -Measures total taste acuity with the patient choosing the appropriate answer ranging from 0=same taste acuity as before treatment to 4=almost complete or complete loss of taste acuity
Time Frame: From baseline through one year after completion of treatment (approximately 15 months)
Reporting Status: Not Posted

10. Other Pre Specified Outcome: Comparison of Quality of Life as Measured by the University of Michigan Xerostomia Index
Description: * Measures impact of salivary gland dysfunction & xerostomia. Scale consists of 15 items covering 4 major domains of oral health-related quality of life: physical functioning, personal/psychological functioning, social functioning, & pain/discomfort issues
  * Patients answer the questions by checking the box that describes the best statement for the past 7 days (not at all, a little, somewhat, quite a bit, very much), 1-5 scale. Higher scores represent greater degree of symptoms. Physical functioning based upon responses to items 1, 6, 10, 12. Pain/discomfort issues based upon responses to items 2, 3, 7, 9. Personal/psychological functioning based upon responses to items 8, 13, 14, 15. Social functioning based upon responses to items 4, 5, 11
  * Captured at baseline, interim assessment (14-42 days post-surgery), Day 1 of radiation, Day 21 after start of radiation, Day 36 after start of radiation, & 6 weeks/4 months/6 months/12 months after completion of adjuvant therapy
Time Frame: From baseline through one year after completion of treatment (approximately 15 months)
Reporting Status: Not Posted

11. Other Pre Specified Outcome: Comparison of Quality of Life as Measured by the MD Anderson Dysphagia Inventory
Description: * Consists of 20 items. Besides a global assessment (a single question), it comprises three subscales: the emotional subscale (8 items), the functional subscale (5 items), and the physical subscale (6 items). The global assessment refers to the individual's swallowing difficulty as it affects one's overall daily routine. The emotional, functional, and physical subscales refer to the individual's affective response to the swallowing disorder, the impact of the disorder on daily activities, and the self-perception of the swallowing difficulties, respectively. Using a five-point scale (1-5), the minimum total score is 20 and the maximum 100
  * Captured at baseline, interim assessment (14-42 days post-surgery), Day 1 of radiation, Day 21 after start of radiation, Day 36 after start of radiation, and 6 weeks/4 months/6 months/12 months after completion of adjuvant therapy
Time Frame: From baseline through one year after completion of treatment (approximately 15 months)
Reporting Status: Not Posted

12. Other Pre Specified Outcome: Comparison of Quality of Life as Measured by the FACT-H&N
Description: * Consists of 27 core items which assess patient function in four domains: Physical, Social/Family, Emotional, and Functional well-being, which is further supplemented by 12 site specific items to assess for head and neck related symptoms. Each item is rated on a 0 to 4 Likert type scale, and then combined to produce subscale scores for each domain, as well as an global QoL score. Higher scores represent better QoL.
  * Captured at baseline, interim assessment (14-42 days post-surgery), Day 1 of radiation, Day 21 after start of radiation, Day 36 after start of radiation, and 6 weeks/4 months/6 months/12 months after completion of adjuvant therapy
Time Frame: From baseline through one year after completion of treatment (approximately 15 months)
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Adverse events were collected from start of treatment through 6 weeks post-end of adjuvant therapy visit.
Description: All-cause mortality, serious adverse events, and other (not including serious) adverse events were not collected for the Not Assigned to an Arm group as these participants did not receive any study treatment.
Arm/Group | Arm 1: POAmCRT | Arm 2: POAmRT | Arm 3: POACRT
All-Cause Mortality (participants affected / at risk) | 0/21 | 0/31 | 0/6
Serious Adverse Events (participants affected / at risk) | 3/21 | 2/31 | 2/6
Other Adverse Events (participants affected / at risk) | 21/21 | 31/31 | 6/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Arm 1: POAmCRT (N=21) | Arm 2: POAmRT (N=31) | Arm 3: POACRT (N=6)
Dehydration (Metabolism and nutrition disorders) | 2 | 0 | 1
Anorexia (Metabolism and nutrition disorders) | 1 | 0 | 0
G-tube pain (Gastrointestinal disorders) | 1 | 0 | 0
Vomiting (Gastrointestinal disorders) | 1 | 0 | 1
Nausea (Gastrointestinal disorders) | 1 | 0 | 1
Oral pain (Gastrointestinal disorders) | 1 | 0 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Chyle leak (Injury, poisoning and procedural complications) | 1 | 0 | 0
Oral hemorrhage (Gastrointestinal disorders) | 0 | 2 | 1
Stoma site infection (Infections and infestations) | 0 | 1 | 0
Fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Hypertension (Vascular disorders) | 0 | 0 | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Atrial flutter (Cardiac disorders) | 0 | 0 | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Arm 1: POAmCRT (N=21) | Arm 2: POAmRT (N=31) | Arm 3: POACRT (N=6)
Anemia (Blood and lymphatic system disorders) | 8 | 14 | 5
Ear pain (Ear and labyrinth disorders) | 1 | 0 | 0
External ear pain (Ear and labyrinth disorders) | 0 | 1 | 0
Hearing impaired (Ear and labyrinth disorders) | 1 | 1 | 1
Tinnitus (Ear and labyrinth disorders) | 1 | 0 | 1
Constipation (Gastrointestinal disorders) | 5 | 5 | 1
Diarrhea (Gastrointestinal disorders) | 2 | 0 | 0
Dry mouth (Gastrointestinal disorders) | 14 | 22 | 4
Dysphagia (Gastrointestinal disorders) | 13 | 27 | 4
Hemorrhoids (Gastrointestinal disorders) | 1 | 0 | 0
Mucositis oral (Gastrointestinal disorders) | 14 | 21 | 4
Nausea (Gastrointestinal disorders) | 9 | 7 | 2
Oral hemmorrhage (Gastrointestinal disorders) | 0 | 0 | 1
Oral pain (Gastrointestinal disorders) | 1 | 4 | 1
Rectal hemorrhage (Gastrointestinal disorders) | 0 | 1 | 0
Vomiting (Gastrointestinal disorders) | 2 | 1 | 1
Chills (General disorders) | 1 | 0 | 1
Edema face (General disorders) | 1 | 4 | 0
Edema limbs (General disorders) | 1 | 0 | 1
Facial pain (General disorders) | 1 | 1 | 0
Fatigue (General disorders) | 12 | 14 | 4
Neck edema (General disorders) | 2 | 0 | 1
Non-cardiac chest pain (General disorders) | 1 | 0 | 0
Pain (General disorders) | 1 | 2 | 1
Sinusitis (Infections and infestations) | 1 | 0 | 0
Dermatitis radiation (Injury, poisoning and procedural complications) | 4 | 5 | 2
Vascular access complication (Injury, poisoning and procedural complications) | 1 | 0 | 0
Activated partial thromboplastin time prolonged (Investigations) | 1 | 1 | 0
Blood bilirubin increased (Investigations) | 0 | 1 | 0
Creatinine increased (Investigations) | 1 | 4 | 2
INR increased (Investigations) | 0 | 1 | 3
Lymphocyte count decreased (Investigations) | 14 | 22 | 4
Neutrophil count decreased (Investigations) | 3 | 0 | 3
Platelet count decreased (Investigations) | 3 | 3 | 3
Weight loss (Investigations) | 16 | 18 | 5
White blood cell decreased (Investigations) | 8 | 7 | 3
Anorexia (Metabolism and nutrition disorders) | 1 | 6 | 2
Dehydration (Metabolism and nutrition disorders) | 0 | 2 | 0
Hypercalcemia (Metabolism and nutrition disorders) | 1 | 0 | 0
Hyperglycemia (Metabolism and nutrition disorders) | 4 | 3 | 2
Hyperkalemia (Metabolism and nutrition disorders) | 3 | 5 | 1
Hypermagnesemia (Metabolism and nutrition disorders) | 1 | 2 | 0
Hypoalbuminemia (Metabolism and nutrition disorders) | 0 | 2 | 1
Hypocalcemia (Metabolism and nutrition disorders) | 1 | 0 | 1
Hypoglycemia (Metabolism and nutrition disorders) | 1 | 1 | 1
Hypokalemia (Metabolism and nutrition disorders) | 0 | 0 | 2
Hypomagnesemia (Metabolism and nutrition disorders) | 1 | 0 | 2
Hyponatremia (Metabolism and nutrition disorders) | 0 | 3 | 2
Hypophosphatemia (Metabolism and nutrition disorders) | 1 | 2 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Muscle weakness right sided (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0
Muscle weakness upper limb (Musculoskeletal and connective tissue disorders) | 0 | 2 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 1 | 3 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 2 | 0
Trismus (Musculoskeletal and connective tissue disorders) | 3 | 0 | 2
Tumor pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Dizziness (Nervous system disorders) | 0 | 0 | 1
Dysgeusia (Nervous system disorders) | 12 | 19 | 2
Headache (Nervous system disorders) | 1 | 0 | 0
Depression (Psychiatric disorders) | 0 | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 2
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 1
Laryngeal inflammation (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Postnasal drip (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Productive cough (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0
Sore throat (Respiratory, thoracic and mediastinal disorders) | 6 | 6 | 0
Voice alteration (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1
Dry skin (Skin and subcutaneous tissue disorders) | 1 | 0 | 1
Rash acneiform (Skin and subcutaneous tissue disorders) | 2 | 0 | 0
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Hematoma (Vascular disorders) | 1 | 0 | 0
Hypertension (Vascular disorders) | 10 | 9 | 2
Lymphedema (Vascular disorders) | 2 | 0 | 0
Superficial thrombophlebitis (Vascular disorders) | 2 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-02-27): https://cdn.clinicaltrials.gov/large-docs/96/NCT03621696/Prot_SAP_001.pdf